CLINICAL TRIAL: NCT01102049
Title: Food-related Differences in Human Metabolite Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 535-ICL-673
Record Dates: First submitted 2010-04-07; First posted 2010-04-12 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — In Situ Hybridization, Fluorescence; Red Meat; Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- self-administered food intake (Experimental): self-administered food intake according to dietary protocol
  Interventions: Dietary Supplement: fish, beef, fruit

INTERVENTIONS:
Dietary Supplement: fish, beef, fruit

SUMMARY:
Many population studies include food questionnaires (recording the normal food intake or the food intake of the study day). This is necessary, because diet is an important lifestyle factor, although food questionnaires are time-consuming and expensive. Moreover, mis-reporting is a very common problem. We therefore seek for a tool to validate food protocol.

The hypothesis is to find biochemical marker for animal protein, fruit intake and grape consumption in urinary metabolic profiles after specific food consumption. Furthermore we want to specify biomarkers for different animal protein sources, fish and beef.

DETAILED DESCRIPTION:
Volunteers are asked to follow a diet plan over the whole course of the study. Every newly introduced food (in this study the dinner on days 2-5) will cause a change in biochemical marker excretion with urine. To monitor the kinetics of biomarker excretion it is necessary to collect urine several times a day; we will ask volunteers to collect the first morning urine, before lunch, before dinner and before going to bed. Urine sampling will start with the first morning urine on day 1 and end with first morning urine on day 7.

As test food, we propose a fruit salad (apples, grapes, orange and grapefruit) on day 2, fish on day 3, grapes on day 4, beef on day 5 and again fish for lunch on day 6.

From day 0 (run-in day) to day 6 the basic diet will always be bread and cheese for breakfast, coffee in the morning, a ham sandwich for lunch, and pasta and tomato sauce for dinner. As beverages only water will be allowed (although wine is permitted on day 4 if the subject wishes but this is not a protocol requirement). The test foods will be consumed in addition to that.

All urine samples will then be analysed using high resolution NMR spectroscopy and mass spectrometry. Mathematical data analyses as well as the visual examinations of the NMR spectra will also be carried out to identify new food biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* male/female
* aged 18-45 years
* non-smoker
* BMI 18-25 kg/m2

Exclusion Criteria:

* regular drug intake
* regular food supplements intake
* antibiotics intake in the last 3 months
* not willing to eat one or more items of the foods listed in the diet plan

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To elucidate urinary biochemical markers for the consumption of fish, beef, fruit salad and grape. | 12 months
  1H NMR metabolic profiles will be acquired for all urine samples. These metabolic profiles contain a wealth of information about metabolites present in urine samples.
  Multivariate mathematical model procedures, such as partial least squares discriminant analysis, will be employed to elucidate metabolic signatures associated to consumption of fish, beef, fruit salad and grape.

SECONDARY OUTCOMES:
To investigate the kinetics of elucidated biomarker excretion over time. | 12 months
  Potential biomarkers (see primary outcome) will be quantified by integrating the NMR resonance and plotted over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Heinzmann SS, Brown IJ, Chan Q, Bictash M, Dumas ME, Kochhar S, Stamler J, Holmes E, Elliott P, Nicholson JK. Metabolic profiling strategy for discovery of nutritional biomarkers: proline betaine as a marker of citrus consumption. Am J Clin Nutr. 2010 Aug;92(2):436-43. doi: 10.3945/ajcn.2010.29672. Epub 2010 Jun 23. PMID 20573794